CLINICAL TRIAL: NCT02505113
Title: Cavernous Transformation of Portal Vein： Etiology, Diagnosis, Management and Prognosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zaibo Jiang, Department of Radiology, The Third Affiliated Hospital, Sun Yat-Sen University, Sun Yat-sen University
Other Study IDs: CTPVDORNO3HSYSU
Record Dates: First submitted 2015-07-16; First posted 2015-07-22 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Portal Vein, Cavernous Transformation Of
Keywords: Portal Vein, Cavernous Transformation Of; Hypertension, Portal
MeSH Terms: conditions — Portal Vein, Cavernous Transformation Of; Hypertension, Portal | interventions — montelukast

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- CTPV without Montelukast: Patients with CTPV do not receive the treatment of Montelukast.
- CTPV treated with Montelukast: Patients with CTPV treated with Montelukast (10mg, q.d., p.o.).
  Interventions: Drug: Montelukast

INTERVENTIONS:
Drug: Montelukast — Montelukast (10mg, q.d., p.o.)
  Groups: CTPV treated with Montelukast

SUMMARY:
To observe the etiology, diagnosis, management and prognosis of cavernous transformation of portal vein.

DETAILED DESCRIPTION:
To observe the etiology, diagnosis, management and prognosis of cavernous transformation of portal vein.

We perform Montelukast (10mg, q.d., p.o.) fot the treatment of symptomatic cavernous transformation of portal vein and to observe the efficacy such as the decrease of the volume of ascites and hydrothorax.

ELIGIBILITY:
Inclusion Criteria:

* All patients with CTPV.

Exclusion Criteria:

* Patients with known severe dysfunction of heart, lung, brain, kidney and other vital organs.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with CTPV
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-10; Primary Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Ascites Volume (mL) | 6 month
  Ascites measured by CT scanning or ultrasound (If the patients had the history of ascites before)
Hydrothorax Volume (mL) | 6 month
  Hydrothorax measured by CT scanning or ultrasound (If the patients had the history of hydrothorax before)

CONTACTS AND LOCATIONS:
Overall Officials: Zaibo Jiang, MD, Study Chair — Sun Yat-sen University
Locations (1):
- Department of Radiology, Guangzhou, Guangdong, China